CLINICAL TRIAL: NCT00230438
Title: A Pilot Study to Develop a Technique for External Beam Radiotherapy After Radical Prostatectomy Based on MRI-Delineation of the Clinical Target Volume
Brief Title: External Beam Radiation Therapy - Target Volume
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 04-0759-CE
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- External Beam Radiation Therapy (Experimental)
  Interventions: Procedure: External Beam Radiotherapy

INTERVENTIONS:
Procedure: External Beam Radiotherapy

SUMMARY:
Delivery of conformal radiation therapy following radical prostatectomy is limited by the inability to define the clinical target volume (CTV). This stems from a poor understanding of patterns of local recurrence and limitations of standard imaging techniques.Magnetic Resonance Imaging (MRI) is a promising modality for imaging the prostatic bed following radical prostatectomy. MRI provides more detailed postoperative anatomy to guide CTV delineation, the ability to document local recurrence patterns, and a method to assess intrafraction prostatic bed motion and deformity to define appropriate planning target volume margins. The aim of this pilot study is to develop a technique for external beam radiation therapy (EBRT) following radical prostatectomy based on MRI-delineation of the CTV. Twenty patients will be enrolled in this pilot, development phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients following radical prostatectomy for prostate adenocarcinoma with one or more of the following adverse features:

pT2 + positive surgical margins ) pT3 ) PSA ≤ 2ng/ml Persistently elevated PSA at 3 months )

* Patients with initially undetectable PSA following prostatectomy for prostate adenocarcinoma with subsequent PSA relapse
* Patients being planned for radiation therapy
* No evidence of distant metastases
* Age ≥ 18 years
* ECOG performance status 0 or 1
* Informed consent

Exclusion Criteria:

* Contraindications to MRI Patients weighing >136 kgs (weight limit for the scanner tables) Patients with pacemakers, cerebral aneurysm clips, shrapnel injury or implantable electronic devices not compatible with MRI.
* Severe claustrophobia
* Inflammatory bowel disease or collagen vascular disease
* Previous colorectal surgery
* Previous pelvic radiotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To develop a technique for MRI-delineation of the clinical target volume (CTV) for EBRT following radical prostatectomy | After data acquisition

SECONDARY OUTCOMES:
To compare the reproducibility of clinical target volume and rectal wall volume delineation on MRI and CT. | After data acquisition
To compare the location of the urethral anastomosis defined on MRI as compared to a fiducial marker placed under TRUS-guidance adjacent to the anastomosis. | After data acquisition
To measure the amount of intrafraction movement and deformity of the prostatic bed and seminal vesicles with current bowel regimen of daily milk of magnesia using cinematic MRI. | After data acquisition
To determine the optimal radiation technique that encompasses the MRI-defined PTV whilst respecting bowel and bladder dose constraints. | After data acquisition
To measure the amount of interfraction movement and deformity of the bladder, rectum, and surgical clips within the operative bed using daily cone-beam CT imaging. | After data acquisition
To explore the utility of IV contrast for the delineation of gross tumor recurrence and normal blood vessels. | After data acquisition

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Menard, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada